CLINICAL TRIAL: NCT00004360
Title: Study of Genotype and Phenotype Expression in Congenital Nephrogenic Diabetes Insipidus
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11929; NU-513
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: Diabetes Insipidus, Nephrogenic
Keywords: diabetes insipidus; endocrine disorders; rare disease
MeSH Terms: conditions — Diabetes Insipidus, Nephrogenic; Diabetes Insipidus; Endocrine System Diseases; Rare Diseases | interventions — Chlorothiazide

INTERVENTIONS:
Drug: chlorothiazide

SUMMARY:
OBJECTIVES:

I. Determine the relationship between genotype variations and clinical phenotype in patients with congenital nephrogenic diabetes insipidus.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: A detailed family history is obtained from all participants. Whenever possible, standard growth curves of affected children are obtained.

Participants then undergo clinical studies of antidiuretic function. A standard fluid deprivation-vasopressin challenge is performed with timed measurements of osmolality, electrolytes, creatinine, and vasopressin. The next day, blood pressure, plasma cyclic AMP, GMP, von Willebrand Factor, Factor VIII, and urine osmolality are measured during a water load desamino-D-arginine vasopressin (dDAVP) infusion test.

Participants with a confirmed diagnosis of congenital diabetes insipidus are then treated with chlorothiazide. Daily urine volume and osmolality are determined before and after therapy. Sodium and fluid are not restricted.

For each family, the entire vasopressin V2 gene of at least 1 affected male, and where possible at least 1 obligate carrier and 1 unaffected brother of a patient is sequenced. In addition, a detailed Xq28 haplotype analysis is done to identify the origin of de novo mutations. If no mutation is found and the disorder is not transmitted in an X-linked mode, both alleles of the gene that codes for aquaporin-II are also sequenced. DNA is collected by mail from as many kindred as possible who do not participate in the clinical studies.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Known or suspected congenital nephrogenic diabetes insipidus
* Clinically and genetically unaffected relatives entered as controls

--Patient Characteristics--

* Age: 6 months to 70 years

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Robertson, Study Chair — Northwestern University

REFERENCES:
- [Background] Bichet DG, Birnbaumer M, Lonergan M, Arthus MF, Rosenthal W, Goodyer P, Nivet H, Benoit S, Giampietro P, Simonetti S, et al. Nature and recurrence of AVPR2 mutations in X-linked nephrogenic diabetes insipidus. Am J Hum Genet. 1994 Aug;55(2):278-86. PMID 8037205
- [Background] Sadeghi H, Robertson GL, Bichet DG, Innamorati G, Birnbaumer M. Biochemical basis of partial nephrogenic diabetes insipidus phenotypes. Mol Endocrinol. 1997 Nov;11(12):1806-13. doi: 10.1210/mend.11.12.0017. PMID 9369448
- [Background] Robertson GL, McLeod JF, Zerbe RL, et al.: Vasopressin function in heritable forms of diabetes insipidus. In: Gross P, Richter D, Robertson GL, eds.: Vasopressin: IV International Vasopressin Conference, May 23-27, 1993, Berlin Germany. Paris: John Libbey Eurotext, 1993, pp 493-503.
- [Background] Wenkert D, Merendino JJ Jr, Shenker A, Thambi N, Robertson GL, Moses AM, Spiegel AM. Novel mutations in the V2 vasopressin receptor gene of patients with X-linked nephrogenic diabetes insipidus. Hum Mol Genet. 1994 Aug;3(8):1429-30. doi: 10.1093/hmg/3.8.1429. No abstract available. PMID 7987330